CLINICAL TRIAL: NCT01127711
Title: Cohort of Swedish Men
Acronym: COSM
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Alicja Wolk, Professor, Karolinska Institutet
Other Study IDs: 1706/2010-631-2
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cancers; Cardiovascular Diseases; Cataract; Gastrointestinal Diseases; Osteoporosis; Fractures
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Cataract; Gastrointestinal Diseases; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Cohort of Swedish Men began in 1997, when all men born between 1918 and 1952 and residing in two counties in central Sweden received a questionnaire including about 350 items concerning diet and other lifestyle factors. A second questionnaire was sent out in 2008-09.

DETAILED DESCRIPTION:
The Cohort of Swedish Men was established in 1997, when all men born between 1918 and 1952 and residing in Västmanland and Örebro counties in central Sweden received a questionnaire concerning diet and other lifestyle factors. Of the 100,303 eligible men, 48,850 (49%) responded to the questionnaire. The questionnaire included items about diet, physical activity, medical history, and lifestyle factors such as cigarette smoking history and use of dietary supplements.

During 2008-09, the exposure information was updated and extended by sending out two new questionnaires - one questionnaire on health including several signs of symptoms, sleeping, social relations etc (2008) and one on diet, dietary supplement use, and lifestyle factors (2009). Majority of questions in the questionnaires have been validated.

Incident cases of cancer are ascertained by record linkages of the study population with the National Swedish Cancer Register and the Regional Cancer Registers. Cardiovascular and other diseases as well as surgeries and causes of death are identified by linkage to the National Inpatient and other registries at the Swedish Board of Health and Welfare. Ascertainment of cancer cases and other diseases is almost 100% complete. Dates of deaths are ascertained through the Swedish Death Register (100% complete), and information on date of moving out of the study area is obtained by linkage with the Swedish Population Register.

ELIGIBILITY:
Inclusion Criteria:

* All men born between 1918 and 1952, living in central Sweden

Exclusion Criteria:

* None

Ages: 45 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men born between 1918 and 1952, living in central Sweden (Örebro and Västmanlands counties)
Sampling Method: Non-Probability Sample
Enrollment: 48850 (Actual)
Dates: Start 1997-09; Primary Completion 1997-12 (Actual)

PRIMARY OUTCOMES:
Prostate cancer | 1997-2010
Pancreatic cancer | 1997-2010
Stomach cancer | 1997-2010
Cataract | 1997-2010
LUTS (Lower urinary tract symptom) | 1997-2010
Cardiovascular Diseases | 1997-2010
Mortality | 1997-2010
Colorectal Cancer | 1997-2010
Bladder cancer | 1997-2010
Fractures, hip fractures | 1997-2014

REFERENCES:
- [Derived] Larsson SC, Drca N, Bjorck M, Back M, Wolk A. Nut consumption and incidence of seven cardiovascular diseases. Heart. 2018 Oct;104(19):1615-1620. doi: 10.1136/heartjnl-2017-312819. Epub 2018 Apr 16. PMID 29661934
- [Derived] Larsson SC, Wallin A, Hakansson N, Stackelberg O, Back M, Wolk A. Type 1 and type 2 diabetes mellitus and incidence of seven cardiovascular diseases. Int J Cardiol. 2018 Jul 1;262:66-70. doi: 10.1016/j.ijcard.2018.03.099. Epub 2018 Mar 24. PMID 29605469
- [Derived] Larsson SC, Wolk A. Potato consumption and risk of cardiovascular disease: 2 prospective cohort studies. Am J Clin Nutr. 2016 Nov;104(5):1245-1252. doi: 10.3945/ajcn.116.142422. Epub 2016 Sep 28. PMID 27680993
- [Derived] Bellavia A, Stilling F, Wolk A. High red meat intake and all-cause cardiovascular and cancer mortality: is the risk modified by fruit and vegetable intake? Am J Clin Nutr. 2016 Oct;104(4):1137-1143. doi: 10.3945/ajcn.116.135335. Epub 2016 Aug 24. PMID 27557655
- [Derived] Xu H, Akesson A, Orsini N, Hakansson N, Wolk A, Carrero JJ. Modest U-Shaped Association between Dietary Acid Load and Risk of All-Cause and Cardiovascular Mortality in Adults. J Nutr. 2016 Aug;146(8):1580-5. doi: 10.3945/jn.116.231019. Epub 2016 Jul 6. PMID 27385761
- [Derived] Larsson SC, Tektonidis TG, Gigante B, Akesson A, Wolk A. Healthy Lifestyle and Risk of Heart Failure: Results From 2 Prospective Cohort Studies. Circ Heart Fail. 2016 Apr;9(4):e002855. doi: 10.1161/CIRCHEARTFAILURE.115.002855. PMID 27072861
- [Derived] Larsson SC, Wallin A, Wolk A. Dietary Approaches to Stop Hypertension Diet and Incidence of Stroke: Results From 2 Prospective Cohorts. Stroke. 2016 Apr;47(4):986-90. doi: 10.1161/STROKEAHA.116.012675. Epub 2016 Feb 11. PMID 26869384
- [Derived] Oskarsson V, Orsini N, Sadr-Azodi O, Wolk A. Fish consumption and risk of non-gallstone-related acute pancreatitis: a prospective cohort study. Am J Clin Nutr. 2015 Jan;101(1):72-8. doi: 10.3945/ajcn.113.076174. Epub 2014 Nov 5. PMID 25527752
- [Derived] Bellavia A, Larsson SC, Bottai M, Wolk A, Orsini N. Differences in survival associated with processed and with nonprocessed red meat consumption. Am J Clin Nutr. 2014 Sep;100(3):924-9. doi: 10.3945/ajcn.114.086249. Epub 2014 Jul 16. PMID 25030780
- [Derived] Bellavia A, Larsson SC, Bottai M, Wolk A, Orsini N. Fruit and vegetable consumption and all-cause mortality: a dose-response analysis. Am J Clin Nutr. 2013 Aug;98(2):454-9. doi: 10.3945/ajcn.112.056119. Epub 2013 Jun 26. PMID 23803880
- [Derived] Larsson SC, Virtamo J, Wolk A. Red meat consumption and risk of stroke in Swedish men. Am J Clin Nutr. 2011 Aug;94(2):417-21. doi: 10.3945/ajcn.111.015115. Epub 2011 Jun 8. PMID 21653800
- See also: Unit of Nutritional Epidemiology — http://ki.se/ki/jsp/polopoly.jsp?l=en&d=20996